CLINICAL TRIAL: NCT00392665
Title: Randomized Study of Bevacizumab/Tarceva and Tarceva/Sulindac in Squamous Cell Carcinoma of the Head and Neck
Brief Title: Bevacizumab/Tarceva and Tarceva/Sulindac in Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Emory University (Other); University of North Carolina, Chapel Hill (Other); Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Lori J. Wirth, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-111
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Keywords: SCCHN; erlotinib; tarceva
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Bevacizumab; Erlotinib Hydrochloride; Sulindac

ARMS (2):
- Erlotinib + Bevacizumab (Active Comparator): erlotinib plus bevacizumab
  Interventions: Drug: Bevacizumab; Drug: erlotinib
- Erlotinib + Sulindac (Active Comparator): erlotinib plus sulindac
  Interventions: Drug: erlotinib; Drug: Sulindac

INTERVENTIONS:
Drug: Bevacizumab — Given intravenously on day one of each 3 week cycle
  Arms: Erlotinib + Bevacizumab
Drug: erlotinib — Given orally once a day
  Other Names: Tarceva
Drug: Sulindac — Given orally twice a day
  Arms: Erlotinib + Sulindac

SUMMARY:
The main purpose of this research study is to collect information to learn how effective erlotinib (tarceva) is in combination with either bevacizumab or sulindac in treating patients with squamous cell carcinoma of the head and neck. Erlotinib and bevacizumab are targeted therapy drugs that can control tumor growth by targeting specific abnormalities sometimes found on cancer cells. Erlotinib targets epidermal growth factor receptor (EGFR), and bevacizumab targets vascular endothelial growth factor (VEGF). Sulindac is a non-steroidal anti-inflammatory drug (NSAID) that can block G protein-coupled receptor which laboratory evidence shows is associated with both cancer cell growth and EGFR activity. The bevacizumab being administered in this study is not a commercially marketed formulation of the drug. Previous research with head and neck cancer suggest that erlotinib alone has some anti-cancer activity. This research study is designed to see how well erlotinib works in combination with bevacizumab or sulindac in head and neck cancer.

DETAILED DESCRIPTION:
* Participants will be randomized to either Arm A: erlotinib plus bevacizumab, or Arm B: erlotinib plus sulindac. Participants will have an equal chance of being placed in any group.
* Medication on Arm A: erlotinib plus bevacizumab: Participants will take erlotinib pills orally once a day. Bevacizumab will be given intravenously on day one of each treatment cycle (each treatment cycle will last three weeks). Urine tests will be performed once every three weeks to test kidney function.
* Medication on Arm B: erlotinib plus sulindac: Participants will take erlotinib pills orally once a day. Sulindac will be taken orally twice a day.
* Physical exams will be performed during each treatment cycle and will include vital signs and general health questions. We will take the participants blood pressure every 2 weeks for the first 6 weeks. After that point, we will take it every 3 weeks or more often if necessary. Blood tests will be performed including chemistry and hematology.
* After every 2 cycles, a repeat CT scan, MRI, and/or PET scan will be performed along with either a chest x-ray or CT scan to ensure that there is no tumor in the participants lungs. We may also do a bone scan if there may be tumor in the participants bones, and abdominal CT scan if there may be tumor in the liver, and a head CT scan or MRI if there may be tumor in the brain.
* After the final treatment the participant will be seen in the clinic to see if they have had any side effects from the drugs within 30 days of stopping the drugs.
* Participants will be in this research study for as long as they are receiving clinical benefits from the study drugs, and do not develop excessive side effects or disease progression. After treatment is discontinued, we will follow the participant closely for 30 days and every 1-2 months after that.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically documented SCCHN, excluding salivary gland primary sites
* 18 years of age or older
* Have evaluable locoregional and/or metastatic disease according to RECIST that is not appropriate for treatment by primary surgical resection or radiotherapy
* Have locoregional and/or metastatic disease that has failed to respond to or relapsed from at least one prior chemotherapy or chemoradiotherapy
* Life expectancy of at least 4 months
* ECOG performance status of 0-2
* Use of effective means of contraception in patients of child-bearing potential

Exclusion Criteria:

* Other malignancy within 5 years except non-melanomatous skin cancer, or carcinoma in situ of the cervix, bladder or head and neck
* Concurrent anticancer therapy other than that of this study
* Treatment with any anticancer drug within 28 days of day 1
* Radiotherapy within 28 days of day 1
* Any unresolved toxicity greater than NCI-CTCAE v 3.0 grade 2 from prior systemic anticancer therapy
* Any prior therapy that targets the ErbB and/or VEGF pathways
* Concurrent therapy with any NSAID
* Known hypersensitivity characterized by acute bronchospasm, urticaria and/or rhinitis to NSAIDs, including aspirin
* Serum creatinine > 1.5 x ULN
* Abnormal LFTs as outlined in protocol
* Blood pressure > 150/100mmHg
* Active unstable angina, or myocardial infarction within 6 months
* NYHA Grade II or greater congestive heart failure
* History of stroke within 6 months
* Clinically significant active peripheral vascular disease
* Absolute neutrophil count < 1000/mm3 or platelets < 100,000/mm3
* Evidence of bleeding diathesis or coagulopathy.
* Tumor encasing the carotid artery, or other major vessel that in the opinion of the investigators is at risk for tumor-related hemorrhage
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspiration or core biopsy within 5 days prior to day 1
* Pregnant or lactating
* History of abdominal fistula or intra-abdominal abscess within 6 months
* History of gastrointestinal ulcer, perforation, or bleeding within 6 months
* Serious non-healing wound or ulcer or active uncontrolled infection
* Bone fracture within 28 days
* Active substance abuse, defined by substance abuse of alcohol, cocaine or intravenous drug use within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Lorch, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib + Bevacizumab | Erlotinib + Sulindac
Started | 18 | 18
Completed | 1 | 3
Not Completed | 17 | 15
Not completed — Death | 16 | 14
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib + Bevacizumab | Erlotinib + Sulindac | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Median (Full Range); unit: years] | 57 [37 to 74] | 57 [37 to 84] | 57 [37 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 17 | 11 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Erlotinib Plus Bevacizumab (Arm A) or Erlotinib Plus Sulindac (Arm B) as Measured by Progression-free Survival.
Description: The primary outcome will be measured by median progression-free survival (PFS), determined by the Kaplan-Meier method for both Arm A and Arm B. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib + Bevacizumab | Erlotinib + Sulindac
Number analyzed (Participants) | 18 | 18
months | 9.38 [4.28 to NA] — the available data does not allow for calculation of an upper bound using the K-M method | 7.01 [2.24 to 11.38]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (complete plus partial response=ORR), as determined by RECIST.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: Two of eighteen patients in both arms had radiographic partial responses, for an overall response rate of 11% for both arms, (95% CI 1.2%, 34.7%). The identical results below are not typos or placeholder values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib + Bevacizumab | Erlotinib + Sulindac
Number analyzed (Participants) | 18 | 18
percentage of participants | 11.1 [1.2 to 34.7] | 11.1 [1.2 to 34.7]

3. Secondary Outcome: Duration of Overall Survival
Description: Median overall survival (OS), determined by the Kaplan-Meier method.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib + Bevacizumab | Erlotinib + Sulindac
Number analyzed (Participants) | 18 | 18
months | 9.38 [4.28 to 14.54] | 8.82 [2.24 to 14.14]

4. Secondary Outcome: Number of Participants With Toxicities According to Severity
Description: Toxicities by Grades 1 or 2 and Grades 3 or 4 in each arm. Grade 4 = life-threatening, Grade 3 = serious, Grade 2 = moderate, Grade 1 = Mild
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib + Bevacizumab | Erlotinib + Sulindac
Number analyzed (Participants) | 18 | 18
Participants
  Fatigue: Grades 1 or 2 | 10 | 8
  Fatigue: Grades 3 or 4 | 0 | 1
  Fatigue: Did not have | 8 | 9
  Rash: Grades 1 or 2 | 14 | 15
  Rash: Grades 3 or 4 | 4 | 1
  Rash: Did not have | 0 | 2
  Diarrhea: Grades 1 or 2 | 8 | 9
  Diarrhea: Grades 3 or 4 | 0 | 0
  Diarrhea: Did not have | 10 | 9
  Hypertension: Grades 1 or 2 | 4 | 0
  Hypertension: Grades 3 or 4 | 0 | 0
  Hypertension: Did not have | 14 | 18
  Oral cavity pain: Grades 1 or 2 | 0 | 2
  Oral cavity pain: Grades 3 or 4 | 0 | 0
  Oral cavity pain: Did not have | 18 | 16
  Dry skin: Grades 1 or 2 | 0 | 2
  Dry skin: Grades 3 or 4 | 0 | 0
  Dry skin: Did not have | 18 | 16
  Hearing problems: Grades 1 or 2 | 0 | 2
  Hearing problems: Grades 3 or 4 | 0 | 0
  Hearing problems: Did not have | 18 | 16
  Dyspepsia: Grades 1 or 2 | 0 | 3
  Dyspepsia: Grades 3 or 4 | 0 | 0
  Dyspepsia: Did not have | 18 | 15
  Dry mouth: Grades 1 or 2 | 0 | 3
  Dry mouth: Grades 3 or 4 | 0 | 0
  Dry mouth: Did not have | 18 | 15
  Constipation: Grades 1 or 2 | 2 | 0
  Constipation: Grades 3 or 4 | 0 | 0
  Constipation: Did not have | 16 | 18
  Anorexia: Grades 1 or 2 | 6 | 0
  Anorexia: Grades 3 or 4 | 0 | 0
  Anorexia: Did not have | 12 | 18
  Dehydration: Grades 1 or 2 | 2 | 0
  Dehydration: Grades 3 or 4 | 0 | 0
  Dehydration: Did not have | 16 | 18
  Dyspnea: Grades 1 or 2 | 2 | 0
  Dyspnea: Grades 3 or 4 | 0 | 0
  Dyspnea: Did not have | 16 | 18
  Mucositis: Grades 1 or 2 | 4 | 2
  Mucositis: Grades 3 or 4 | 0 | 0
  Mucositis: Did not have | 14 | 16
  Neuropathy-sensory: Grades 1 or 2 | 0 | 2
  Neuropathy-sensory: Grades 3 or 4 | 0 | 0
  Neuropathy-sensory: Did not have | 18 | 16
  Hemmorrhage: Grades 1 or 2 | 8 | 0
  Hemmorrhage: Grades 3 or 4 | 0 | 0
  Hemmorrhage: Did not have | 10 | 18
  Nausea: Grades 1 or 2 | 4 | 2
  Nausea: Grades 3 or 4 | 0 | 0
  Nausea: Did not have | 14 | 16
  Vomiting: Grades 1 or 2 | 2 | 0
  Vomiting: Grades 3 or 4 | 0 | 0
  Vomiting: Did not have | 16 | 18
  Insomnia: Grades 1 or 2 | 2 | 0
  Insomnia: Grades 3 or 4 | 0 | 0
  Insomnia: Did not have | 16 | 18
  Pruritus: Grades 1 or 2 | 0 | 2
  Pruritus: Grades 3 or 4 | 0 | 0
  Pruritus: Did not have | 18 | 16
  Hypomagnesemia: Grades 1 or 2 | 2 | 2
  Hypomagnesemia: Grades 3 or 4 | 0 | 0
  Hypomagnesemia: Did not have | 16 | 16

ADVERSE EVENTS:
Arm/Group | Erlotinib + Bevacizumab | Erlotinib + Sulindac
Serious Adverse Events (participants affected / at risk) | 4/18 | 5/18
Other Adverse Events (participants affected / at risk) | 18/18 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib + Bevacizumab (N=18) | Erlotinib + Sulindac (N=18)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vascular access-Thrombosis/embolism (Vascular disorders) | 0 (0) | 1 (1) — fatal, unlikely related
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nonneuropathic right-side muscle weak (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib + Bevacizumab (N=18) | Erlotinib + Sulindac (N=18)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 13 (24) | 11 (18)
Fatigue (General disorders) | 13 (21) | 12 (19)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 7 (10) | 8 (10)
Nausea (Gastrointestinal disorders) | 7 (9) | 5 (8)
Dry mouth (Gastrointestinal disorders) | 7 (8) | 8 (14)
Dysphagia (Gastrointestinal disorders) | 6 (7) | 5 (6)
Constipation (Gastrointestinal disorders) | 5 (10) | 3 (3)
Oral cavity- pain (General disorders) | 5 (9) | 2 (5)
Hypertension (Cardiac disorders) | 5 (7) | 0 (0)
Head/headache (General disorders) | 5 (5) | 1 (1)
Anorexia (Gastrointestinal disorders) | 4 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4)
Hemorrhage-other (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (5) | 3 (3)
Pain-other (General disorders) | 4 (5) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 4 (4) | 2 (4)
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 4 (4) | 1 (2)
Nose- hemorrhage (Blood and lymphatic system disorders) | 4 (4) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Neuropathy-sensory (Nervous system disorders) | 3 (4) | 4 (6)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Dehydration (Gastrointestinal disorders) | 3 (3) | 1 (2)
Rigors/chills (General disorders) | 3 (3) | 1 (1)
Skin-other (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (3)
Throat/pharynx/larynx- pain (General disorders) | 2 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
GI-other (Gastrointestinal disorders) | 2 (3) | 2 (3)
Anxiety (Nervous system disorders) | 2 (2) | 1 (3)
AST- SGOT (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Back- pain (General disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Edema head and neck (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Edema limb (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Infection-other (Infections and infestations) | 2 (2) | 1 (1)
Insomnia (General disorders) | 2 (2) | 1 (1)
Ocular-other (Eye disorders) | 2 (2) | 1 (1)
Pain NOS (General disorders) | 2 (2) | 5 (6)
Sweating (General disorders) | 2 (2) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (2) | 3 (4)
Neck- pain (General disorders) | 1 (2) | 2 (3)
Salivary (Gastrointestinal disorders) | 1 (2) | 2 (2)
Abdomen- pain (General disorders) | 1 (1) | 1 (1)
ALT- SGPT (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bilirubin (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Chelitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Depression (Nervous system disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (4)
Hyopthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Renal/GU-other (Renal and urinary disorders) | 1 (1) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hearing-other (Ear and labyrinth disorders) | 0 (0) | 3 (4)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No